CLINICAL TRIAL: NCT01945541
Title: Body Composition Monitoring for Determination of the Fluid Status in Patients Undergoing General Anesthesia
Brief Title: Body Composition Monitoring(BCM) for Determination of the Fluid Status in Patients Undergoing General Anesthesia
Acronym: BCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Kabon, PD. MD., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2059/2012
Record Dates: First submitted 2013-08-31; First posted 2013-09-18 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Fluid Overload
Keywords: Intraoperative Fluid Administration; Body Composition Measurement
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard fluid management (No Intervention): postoperative BMC measurements
- body composition monitoring preoperative (Active Comparator): pre and postoperative BCM measurements
  Interventions: Device: Body Composition Monitoring

INTERVENTIONS:
Device: Body Composition Monitoring — Pre- and postoperative measurements of body composition (intracellular and extracellular water content)via bioimpedance spectroscopy
  Other Names: Fresenius Healthcare Germany
  Arms: body composition monitoring preoperative

SUMMARY:
The purpose of this study is to evaluate a recently developed device, which measures body composition (i.e. the water content of the body) in the perioperative setting. Specifically the investigators will test the hypothesis, that extracellular water content after surgery correlates to the amount of intraoperative infusion and positive fluid balance. Furthermore the investigators will test, if preoperative evaluation of body water helps to determine intraoperative fluid requirements and to guide fluid administration.

DETAILED DESCRIPTION:
Patients undergoing anesthesia and surgery receive intravenous fluids during the procedure. The amount of administered fluid depends on the type of surgery, cardiovascular stability and intraoperative losses like hemorrhage. Fluid overload as well as hypohydration might be detrimental and might adversely effect outcome after surgery. Specifically overhydration results in significant weight gain, tissue edema and increased morbidity. Technically assisted assessment of volume status before surgery may be useful to direct intraoperative fluid administration and to prevent postoperative volume overload. As a prerequisite the investigators will test a recently developed whole-body bioimpedance spectroscopy device to determine the pre-to postoperative fluid distribution. This body composition monitor (BCM, Fresenius Medical Care, Germany) separates between extracellular and intracellular fluid volume non-invasively by applying a frequency sweep from 3-1000 kilohertz through the entire patient via electrodes placed on the wrist and ankle.

The investigators will test the hypothesis that

1. the amount of administered fluid correlates with the amount of overhydration measured postoperatively.
2. that preoperative BCM measurements and thus information about the preoperative hydration state might help to guide fluidmanagement and to reduce the amount of over/ hypohydration postoperatively.

ELIGIBILITY:
Inclusion Criteria:

18-80 Years

Exclusion Criteria:

liver, heart, kidney failure, patients with pacemaker

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-08-24 (Actual)

PRIMARY OUTCOMES:
Postoperative overhydration in liter measured by Body Composition Monitor | Measurements will be performed immediatley before and after surgery. The expected time frame will thus be 2-4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kabon, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria